CLINICAL TRIAL: NCT05903430
Title: A Feasibility Study of MRI Guided Stereotactic Ablative Radiotherapy
Brief Title: A Feasibility Study of MRI Guided Stereotactic Ablative Radiotherapy (MIDSECTION)
Acronym: MIDSECTION
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTsp194
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Cancer; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The optional biospecimens collected and stored from patients will include some or all of the following; tissue in the form of a diagnostic block (likely Formalin Fixed Paraffin Embedded FFPE), whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine if the investigators are able to deliver highly focused, intense radiation to tumours in the abdominal region or chest cavity whilst limiting the dose to surrounding organs using a high field strength MR-Linac.

DETAILED DESCRIPTION:
Stereotactic Ablative Radiotherapy (SABR) for tumours in the thorax and abdomen is becoming the standard of care for patients with small, localised disease. Recent publications and guidelines provide evidence for safe, effective treatment prescriptions in most of these tumour sites. However this guidance is based on the use of x-ray based guidance systems, without the use of functional imaging or real-time adaptation. To investigate the potential benefits of MRI-guided SABR, including superior at-treatment imaging, gating, real-time adaptation and the integration of functional or biological information, the investigators propose to undertake MR-guided SABR using established guidance. In doing this the investigators will be able to evaluate the patient experience (for example the MR Linac is considerably noisier than a standard treatment machine); the investigators will be able to acquire images (with no additional radiation) to interrogate motion, and deformations in real-time to assess whether or not real time adaptations would benefit the patient experience and/or outcomes; the investigators will be able to compare the outcomes of the patients treated on a machine with superior imaging to those undergoing the same (or similar) treatment on standard machines using the UKCAT database; the investigators will be able (should participants choose to give consent) to acquire research images interrogating tumour and normal tissue physiology/biology and determine if and how this information may be able to improve treatments and/or predict response. For these reasons it is important to make this change in practice (from x-ray guided SABR to MRI-guided SABR) within the confines of an observational clinical study.

ELIGIBILITY:
Inclusion criteria:

1. Have no MRI contra-indications.
2. Eligible for abdominal SABR in accordance with the NHSE SABR Consortium Guidelines or eligible for central lung SABR in accordance with RTOG Guidelines.
3. Be able to give informed consent.
4. Anticipated life-expectancy > 6 months.
5. Not more than 3 oligmetastatic sites treated in total per patients.
6. Performance status ≤ 2.
7. Willing to attend follow-up and have details collected on prospective basis for a minimum of 1 year.

Exclusion criteria:

1. Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form.
2. Unable to tolerate MRI scans.
3. Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator make it undesirable for the patient to participate in the study.
4. Any evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator, make it undesirable for the patient to participate in the study.
5. Any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Either patient with abdominal cancer or centrally located lung cancer eligible for SABR
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
> 85% success in delivery and completion of radiotherapy to patients recruited on protocol | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No